CLINICAL TRIAL: NCT01812109
Title: Near-Infrared Spectroscopy for Pediatric Acute Scrotum and Testicular Torsion
Acronym: NIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Linda A Baker, Professor of Urology, Director of Pediatric Urology Research, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 102010-133; 1R21DK092654-01A1 (NIH)
Record Dates: First submitted 2013-01-24; First posted 2013-03-15 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Acute Scrotum; Testicular Torsion
Keywords: Testicular Torsion
MeSH Terms: conditions — Spermatic Cord Torsion

STUDY DESIGN:
Intervention Model Description: Those that accept study participation after informed consent will receive standard of care therapy for the acute scrotum and will be evaluated by NIRS. The NIRS measurements will not bias the treatments performed or not performed on the study patients, permitting standard of care treatment unbiased. The clinical data will be collected prospectively for each patient utilizing REDCap Data Collection Management and stored in the REDCap databases and the photographic database. Photographs will be taken of the scrotum. In addition, select participants will be asked if they will allow us to videotape the NIRS measurements.
Masking Description: The probe will be laid on the exposed testis (intraoperative testicular tissue). Each measurement is painless and takes <15 seconds each. The NIRS probe will be placed on the anterior testis to obtain the three sets of three measurements. Thus, the unaffected testis will serve as the patient's own control. NIRS #2-4 will not delay detorsion of the affected testis. Surgeons will be blinded to these NIRS results, thus the decision during the operation will not be affected.
  All participants' NIRS results will be blinded to the surgeons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hutchison Technologies Inspectra StO2 NIRS (Experimental): Hutchison Technologies Inspectra StO2 SpotCheck Near-Infrared Spectroscopy (NIRS) evaluation of acute scrotum per protocol
  Interventions: Device: Hutchison Technologies Inspectra StO2 SpotCheck Near-Infrared Spectroscopy

INTERVENTIONS:
Device: Hutchison Technologies Inspectra StO2 SpotCheck Near-Infrared Spectroscopy — Device: Near-Infrared Spectroscopy Transscrotal NIRS is a series of 6 transcutaneous scrotal measurements, 3 on both left/right. Each measurement is completely non-invasive, painless and takes ~15 seconds each. Thus, no sedation or supplemental analgesia is needed for NIRS. The NIRS probe will be placed on the anterior, lateral and posterior scrotum on the left/right sides, immediately overlying and parallel to the long axis of the testis but on the skin to obtain the 6 total measurements. The unaffected testis will serve as the patient's own control. Study coordinators will be performing the ER transscrotal NIRS testing. For uniformity, all will be trained for testicular probe placement methods. NIRS will not delay the gray scale/color Doppler testicular US or surgery.

SUMMARY:
Testicular torsion is the spontaneous twisting of the testis and its blood vessels, resulting in acute pain, vascular compromise and death of the testicle if unrelieved quickly. In this study, investigators will test a near-infrared spectroscopy (NIRS) device that rapidly and non-invasively measures deep tissue oxygen saturation.

DETAILED DESCRIPTION:
The main goal of this prospective, non-randomized pilot study is to assess the utility of NIRS for the clinical diagnosis of the acute scrotum and testicular torsion. The sensitivity and specificity of NIRS for testicular torsion will be defined relative to surgical exploration, scrotal Doppler/B-mode ultrasound, and clinical follow-up. Last, we will assess the utility of intraoperative and postoperative NIRS for predicting testicular viability after testicular detorsion. To achieve this, standard care will be provided for all patients and at two or five time points NIRS measurements will be obtained privately so standard care is not biased by NIRS data. Outcome variables will include NIRS StO2 ( percent oxygen saturation) measurements, torsion status (yes/no), ultrasound parameters (testicular size, volume, echogenicity, presence/absence of Doppler flow, whirlpool sign, hydrocele, scrotal wall thickness), TWIST score variables, duration of pain, and duration of torsion. Study endpoints will include early withdrawal, screen failures, orchiectomy for torsion, and 1-2 week or 3 month post-surgical follow-up (see Figure 1). In this 5 year single center study, the maximum number of local subjects to be consented will be 750 subjects. No existing charts will be used in this prospective study.

Patients with acute scrotum will be evaluated by history, physical examination, and urinalysis per standard of care by staff in the ER, pediatric urology or pediatric surgery. At the surgeon's discretion, either a scrotal Doppler/B-mode ultrasound or emergent surgical exploration will be planned as the next step per standard of care. While waiting for preparation of either the scrotal Doppler/B-mode ultrasound or emergent surgical exploration, the patient and guardian will be informed and invited for study participation. If they agree to participate, they will be given a Fitzpatrick Skin Type (FST) Survey. This survey is a classification scale that was created in 1975 for predicting skin reactivity in PUVA (Psoralen plus ultraviolet A) photochemotherapy. [20] This survey asks the subject to grade his tendency to burn and ability to tan respectively within 24 hours and 7 days after the first un-protected sun-exposure in the early summer. There are four possible answers for "white"-skinned persons (skin type I, II, II, IV). Brown skin classification is skin type V and black skin classification is skin type VI. In the event that the survey has been missed, we will mail a survey to the patient/guardian with a pre-stamped and addressed return envelope. [20] Those that refuse study participation will receive standard of care treatment for the acute scrotum.

Those that accept study participation after informed consent will receive standard of care therapy for the acute scrotum and will be evaluated by NIRS. The NIRS measurements will not bias the treatments performed or not performed on the study patients, permitting standard of care treatment unbiased. The clinical data will be collected prospectively for each patient utilizing REDCap Data Collection Management and stored in the REDCap databases and the photographic database. Photographs will be taken of the scrotum. In addition, select participants will be asked if they will allow us to videotape the NIRS measurements.

At the surgeon's decision and discretion, either a scrotal Doppler/B-mode ultrasound or emergent surgical exploration will be planned as the next step per standard of care. While waiting for this to occur, the NIRS #1 measurement will be obtained. NIRS #1 is a series of 6 transcutaneous scrotal measurements, three on the left and three on the right. Each measurement is completely non-invasive, painless and takes <15 seconds each. Thus, no sedation or supplemental analgesia will be needed for NIRS. The NIRS probe will be placed on the anterior scrotum on the left and right sides, immediately overlying the testis but on the skin, to obtain the six total measurements. Thus, the unaffected testis will serve as the patient's own control. NIRS #1 will not delay the scrotal Doppler/B-mode ultrasound or emergent surgical exploration.

If the surgeon decides against surgical exploration, then standard care for the other causes of acute scrotum will be provided and the diagnosis will be no testicular torsion. The patient will be discharged home with a standard care follow-up in approximately two weeks in an outpatient urology clinic appointment. The subject will be given a NIRS Daily Diary to take home with them and record a five-day history of pain and recovery course. They will be asked to bring this back at the two week follow-up visit.

If the scrotal Doppler/B-mode ultrasound identifies testicular torsion or if the surgeon feels emergent surgical exploration is indicated, then emergent surgical exploration will be performed. Photographs of the scrotum will be obtained, as well as select patients to be consented for videotaping of the NIRS measurements At surgery under general anesthesia per standard care, NIRS #2-4 will be performed. NIRS #2-4 is a series of 18 testicular tissue measurements, nine on the affected testis and nine on the unaffected testis. Each testis will receive nine measurements, three thru the skin and six directly on the exposed testis (three prior to untwisting and three 5 minutes after untwisting). The probe will be laid on the exposed testis (intraoperative testicular tissue). Each measurement is painless and takes <15 seconds each. The NIRS probe will be placed on the anterior testis to obtain the three sets of three measurements. Thus, the unaffected testis will serve as the patient's own control. NIRS #2-4 will not delay detorsion of the affected testis. Surgeons will be blinded to these NIRS results, thus the decision during the operation will not be affected.

In addition, using a standardized color wheel we have created, the surgeon will be asked to describe the color of the testis at the time of initial exposure and at 5 minutes after detorsion.

If testicular torsion is found and the torsed testis is nonviable after detorsion, the orchiectomy with contralateral orchiopexy will be performed per surgeon's decision. The patient will be discharged home and will reach study endpoint.

If testicular torsion is found and the torsed testis is viable after detorsion, then bilateral orchiopexy will be performed. One hour after the NIRS #2-4 measurements were completed, NIRS #5 will be performed using the method described for NIRS #1 only on postsurgical patients that underwent bilateral orchiopexy for testicular salvage.

At the time of discharge home, the subject will be given a NIRS Daily Diary to take home with them and record a five-day history of pain and recovery course. They will be asked to bring this back at the two week follow-up visit.

A phone interview will take place at day 5 to assess their postoperative pain course. A telephone script will be utilized if the patients fail to follow-up with the urology clinic. We will conduct this brief telephone interview with the parents/guardians as a means of follow-up.

1-2 weeks later, non-surgical patients and surgical patients having bilateral orchiopexy will return for an outpatient urology clinic evaluation of ~1 hour duration.

1. After standard care clinical evaluation, if the diagnosis is still no testicular torsion, then the patient is discharged home and reaches study endpoint.
2. After standard care clinical evaluation, if there is a clinical concern over testicular viability (missed testicular torsion), then a repeat standard care scrotal Doppler/B-mode ultrasound will be obtained immediately and NIRS #6 will be performed using the method described for NIRS #1. The patient will be categorized as torsion or no torsion based on clinical findings and reaches study endpoint. In addition, photographs of the scrotum and possible selected videotaping will be performed.
3. As per standard of care, if testicular torsion was present and the testis underwent detorsion with orchiopexy, then NIRS #6 will be performed using the method described for NIRS #1. At 3 months post-operatively, a scrotal Doppler/B-Mode Ultrasound will be obtained to assess testicular volume and dimensions, which is standard of care follow-up after orchiopexy. The affected testis will be categorized as normal, <20% testicular volume loss, 20-50% volume loss, or >50% volume loss based on ultrasound parameters. At that ~1 hour visit, NIRS #7 will be performed using the method described for NIRS #1, photographs of the scrotum and possible selected videotaping will be performed. At that time, the patient reaches study endpoint.

If the patient does not return at either the designated 1-2 weeks or three month follow-up outpatient urology clinic evaluation, then the PI and/or research nurse coordinator will telephone the guardian to encourage return to clinic and for verbal status report on the child's clinical state.

Thus, the total number of study visits, including the presenting emergency visit, is three (Emergency, 1-2 weeks post-operatively, and 3 months post-operatively). No medications will be administered in this study. No blood or tissue will be collected and no radiation exposure or questionnaires will be given. No subjects will be responsible for any research-related costs however; they will be responsible for standard care costs. At the end of the study, standard care will be turned over to the primary care physician or pediatric urologist if needed. No sub-study procedures will be performed.

ELIGIBILITY:
Inclusion Criteria:

Males one month to 21 years of age with:

Painful acute scrotum or testis OR Abdominal pain (+/- nausea, vomiting) and waddling gait ("cowboy shuffle") from painful scrotum.

Exclusion Criteria:

Males with:

Synchronous bilateral testicular torsion History of known testicular or scrotal surgery Current hernia or painless hydrocele Current obvious scrotal bug bites History of chronic respiratory, hematological or vascular problems that will affect total body tissue oxygenation levels (Home oxygen).

Ages: 1 Month to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 154 (Actual)
Dates: Start 2011-03-24 (Actual); Primary Completion 2015-03-25 (Actual); Study Completion 2015-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Baker, MD, Principal Investigator — University of Texas
Locations (1):
- Children's Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Background] DaJusta DG, Granberg CF, Villanueva C, Baker LA. Contemporary review of testicular torsion: new concepts, emerging technologies and potential therapeutics. J Pediatr Urol. 2013 Dec;9(6 Pt A):723-30. doi: 10.1016/j.jpurol.2012.08.012. Epub 2012 Oct 6. PMID 23044376
- [Result] Sheth KR, Keays M, Grimsby GM, Granberg CF, Menon VS, DaJusta DG, Ostrov L, Hill M, Sanchez E, Kuppermann D, Harrison CB, Jacobs MA, Huang R, Burgu B, Hennes H, Schlomer BJ, Baker LA. Diagnosing Testicular Torsion before Urological Consultation and Imaging: Validation of the TWIST Score. J Urol. 2016 Jun;195(6):1870-6. doi: 10.1016/j.juro.2016.01.101. Epub 2016 Feb 2. PMID 26835833
- [Result] Schlomer BJ, Keays MA, Grimsby GM, Granberg CF, DaJusta DG, Menon VS, Ostrov L, Sheth KR, Hill M, Sanchez EJ, Harrison CB, Jacobs MA, Huang R, Burgu B, Hennes H, Baker LA. Transscrotal Near Infrared Spectroscopy as a Diagnostic Test for Testis Torsion in Pediatric Acute Scrotum: A Prospective Comparison to Gold Standard Diagnostic Test Study. J Urol. 2017 Sep;198(3):694-701. doi: 10.1016/j.juro.2017.03.134. Epub 2017 Apr 6. PMID 28392394
- [Result] Grimsby GM, Schlomer BJ, Menon VS, Ostrov L, Keays M, Sheth KR, Villanueva C, Granberg C, Dajusta D, Hill M, Sanchez E, Harrison CB, Jacobs MA, Burgu B, Hennes H, Baker LA. Prospective Evaluation of Predictors of Testis Atrophy After Surgery for Testis Torsion in Children. Urology. 2018 Jun;116:150-155. doi: 10.1016/j.urology.2018.03.009. Epub 2018 Mar 20. PMID 29572055

RESULTS

PARTICIPANT FLOW:
Groups:
- NIRS: There is only 1 group in this non randomized pilot study. Those patients with acute scrotum defined as painful scrotum or testes, abdominal pain +/- nausea and vomiting, waddling gain (cowboy shuffle) .
Period: Overall Study
Arm/Group | NIRS
Started | 154
With Torsion | 36
Without Torsion | 85
Completed | 121
Not Completed | 33
Not completed — research personnel delay | 16
Not completed — NIRS Unattainable | 17

BASELINE CHARACTERISTICS:
Population: 17 participants were excluded from the analysis as the NIRS reading could not be obtained.
Arm/Group | NIRS
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 121
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  Hispanic | 79
  Black | 15
  Asian | 1
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Median NIRS Delta %StO2
Description: Testicular tissue percent oxygen saturation (%StO2) is measured by transscrotal near infrared spectroscopy (NIRS). This is similar to the PulseOx machine that is usually used when we go for a regular doctor visit.
  NIRS measurements were obtained with Hutchison Technology InSpectra StO2 Spot Check Device (Model 300) with thenar clip probe (Model 1315, modified by clip removal).
  Measurements were done at 1, 5 and 10 seconds to account for interassay variability, which is expected to be less than 3 %StO2. The average of the 3 readings was defined as the NIRS %StO2 reading for that testis. The NIRS readings in the affected testis were normalized to the contralateral normal testis to formulate a NIRS delta %StO2 (%StO2 of unaffected testis and %StO2 of affected testis). If the affected testis had lower %StO2 readings than the contralateral normal testis, NIRS delta %StO2 would be positive.
Time Frame: Done at 1, 5 and 10 seconds
Population: Here we are reporting Median NIRS delta %StO2 with Torsion and without torsion.
Measure: Median (Inter-Quartile Range); unit: percentage of StO2
Arm/Group | Hutchison Technologies Inspectra StO2 NIRS
Number analyzed (Participants) | 121
percentage of StO2
  Torsion: number analyzed (Participants) | 36
  Torsion | 2.0 [-4.2 to 9.8]
  No Torsion: number analyzed (Participants) | 85
  No Torsion | -1.7 [-8.7 to 2.0]

ADVERSE EVENTS:
Time Frame: Baseline upto 2weeks post -op.
Description: No Adverse events occurred in this study.
Arm/Group | Hutchison Technologies Inspectra StO2 NIRS
All-Cause Mortality (participants affected / at risk) | 0/154
Serious Adverse Events (participants affected / at risk) | 0/154
Other Adverse Events (participants affected / at risk) | 0/154

LIMITATIONS AND CAVEATS:
Different NIRS probes may be needed for prepubertal vs postpubertal testis and further research is needed to optimize NIRS device configuration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No